CLINICAL TRIAL: NCT06619782
Title: Practice Facilitation to Enhance Implementation of a Pediatric Suicide Prevention Pathway
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 23-2155; R34MH132832 (NIH)
Record Dates: First submitted 2024-09-20; First posted 2024-10-01 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Suicide Prevention
Keywords: suicide prevention; pediatric primary care; practice facilitation
MeSH Terms: conditions — Suicide Prevention

STUDY DESIGN:
Intervention Model Description: The intervention involves training and implementation of the NIMH suicide prevention pathway in pediatric primary care and family medicine practices
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Practice Facilitation (Experimental): Practice facilitation is added to training in the suicide prevention pathway in primary care to provide implementation support for integrating the pathway into routine care
  Interventions: Other: Practice Facilitation; Other: Training in National Institute of Mental Health Youth Suicide Prevention Pathway
- Training Only (Active Comparator): Primary care practices are trained in the National Institute of Mental Health (NIMH) youth suicide prevention pathway without practice facilitation
  Interventions: Other: Training in National Institute of Mental Health Youth Suicide Prevention Pathway

INTERVENTIONS:
Other: Practice Facilitation — Practice facilitation (PF) is a supplemental support to increase competence and and adoption of the National Institute of Mental Health (NIMH) youth suicide prevention. pathway in primary care. Practices will receive 6 months of PF which involves clinic- and provider- level data review and adoption data for the 5 components of the prevention pathway, clinical coaching around implementing the different components , logistical coaching in identifying multilevel contextual barriers to implementation and strategies to overcome them
  Arms: Practice Facilitation
Other: Training in National Institute of Mental Health Youth Suicide Prevention Pathway — Training in the National Institute of Mental Health (NIMH) Youth Suicide Prevention Pathway involves a 2-hour in-person presentation created in consultation with NIMH, Zero Suicide and Substance Abuse and Mental Health Services Administration. It is delivered by a licensed professional counselor with content expertise to all primary care practice personnel involved in the prevention pathway. The first hour focuses on conducting Ask Suicide Screening Questions (ASQ) screening, identifying risk/protective factors, identifying warning signs and conducting a brief suicide safety assessment. The second hour covers safety planning, lethal means safety, behavioral health referrals and arranging follow-up. Didactic and interactive methods are used, including group discussion, activities, videos and case vignettes

SUMMARY:
Suicide in youth is rapidly growing to where it is the second leading cause of death across the United States. Use of available tools have shown the potential to boost primary care providers' (PCPs) detection of suicide risk and confidence and knowledge around addressing it; however, ways that work to address clinic and provider barriers that influence the ongoing implementation of a pathway to manage at-risk patients remain under researched. The proposed study will assess the impact of the investigators Facilitated Suicide Prevention program--which provides support to assist practices in integrating screening, assessment, data analysis and management procedures into routine care through feedback and coaching--on clinic use of the suicide prevention pathway and youth suicide.

The project hypothesizes that compared to PCPs in Training Only (TO) practices, those in TO+Practice Facilitation (PF) may rate the care pathway as more able to be carried out and acceptable; demonstrate greater use of the pathway components (screening, risk assessment, safety planning, lethal means safety counseling, referrals and follow-up); demonstrate higher levels of use of the pathway suicide prevention skills ; and report higher levels of confidence putting the care pathway into use.

Also we predict that, compared to youth who screen positive for suicide risk and are followed by PCPs in TO practices, those who screen positive and are followed by PCPs in TO+PF practices will be less likely to attempt suicide during the next six months; less likely to have suicidal ideation during the next 6 months; more likely to see a behavioral health provider during the next 6 months; and less likely to be sent to Emergency Departments during the next 6 months .

DETAILED DESCRIPTION:
Suicide is a leading cause of death in youth across the United States. Approximately 80% of youth who die by suicide interface with the medical system in the year preceding their death. Primary care practices (PCPs) serving youth are well positioned to detect patients at risk for suicide and intervene, and widely accessible toolkits are available for practices to use. However, effective ways to impact providers' skills in actually carrying out a clinical pathway to manage at-risk patients remain under researched. Indeed, training without applied practice and support is likely not enough to significantly have an effect on these skills in the long term and less likely to improve patient outcomes. Practice facilitation is a powerful way to transform clinical practice, develop provider skills, and improve patient outcomes. The investigators train PCPs in the National Institute of Mental Health (NIMH) youth suicide prevention care pathway and, in addition, assists them in integrating the pathway into routine care with feedback and support through practice facilitation and data collection. However, there is limited evidence for the effects of supports, such as practice facilitation or coaching, on primary care providers' use of and skills in suicide risk assessment and management. Thus, guided by the combined Reach, Effectiveness, Adoption, Implementation, Maintenance (RE-AIM)/Practical Robust Implementation and Sustainability (PRISM) framework, this study will compare the impact of practice facilitation added to suicide prevention training based on the NIMH youth suicide prevention care pathway (TO+PF) versus training only (TO). In this study, Pediatric and Family Medicine practices in collaborating practice-based research networks will be assigned to TO+PF or to TO. Providers in TO+PF clinics will receive practice facilitation for 6 months, involving monthly individual check-ins which include: 1) clinic- and provider-level data review of use data for the five components of the NIMH youth suicide prevention care pathway, 2) clinical coaching around implementing the different components of the pathway, and 3) coaching in identifying barriers to use and strategies to overcome them. At the clinic/provider level, the feasibility, acceptability, effectiveness, adoption, fidelity, use and barriers will be measured. At the patient level, youth assessed at intermediate or high risk and their family will be followed for 6 months following, with data collected on attempted suicides and suicide ideation as well as emergency room and behavioral health provider visits. The outcomes will provide preliminary support for a subsequent larger. study of the suicide prevention pathway, assessing its use, impact, and sustainability, with the goal of promoting broad use in a variety of clinic contexts.

ELIGIBILITY:
Inclusion Criteria:

Youth

* between the ages of 12 and 24 years
* present to a participating PCP and practice for a well visit
* receive a positive ASQ screen during their well visit. Providers
* All staff in enrolled Primary Care practices (e.g., physicians, physician assistants nurses, administrative staff) will be eligible to participate and complete relevant measures.

Exclusion Criteria:

Youth

* Over 24 years
* Do not receive a positive ASQ screen at well visit.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Ask Suicide Screening Questions | At enrollment (baseline) and 6 months (study completion)
  A set of four brief suicide screening questions that takes 20 seconds to administer. A validated tool that is approved for use by the Joint Commission for all ages
Suicidal Ideation Questionnaire | At enrollment (baseline) and 6 months (study completion)
  The Suicidal Ideation Questionnaire (SIQ) assesses the frequency of suicidal ideation.The SIQ consists of 30 items and is appropriate for students in Grades 10-12. The Suicidal Ideation Questionnaire-Junior (SIQ-JR) consists of 15 items and is designed for students in Grades 7-9, consists of a subset of items from the original SIQ. For both the SIQ and SIQ-Jr, the stem indicates "Listed below are a number of sentences about thoughts that people sometimes have. Each item has 7 response options ranging from 0 ("I never had this thought") to 6 ("almost every day"). Scoring is done by summing the item response scores for a range of 0 to 180 for the SIQ and 0 to 90 for the SIQ-JR, with higher scores indicating the presence of more symptomatology.
Patient Health Questionnaire-9 | At enrollment (baseline) and 6 months (study completion)
  A 9- item measure that assesses the severity of depressive disorders and episodes (or clinically significant symptoms of depressive disorders and episodes) in children ages 11-17. It was adapted from Patient Health Questionnaire-9 modified for Adolescents (PHQ-A]). Possible range of scores is 0 to 27, with the higher scores indicating the presence of more symptomatology. Total scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively.
Center for Epidemiological Studies Depression Scale (CES-D) | At enrollment (baseline) and 6 months (study completion)
  Center for Epidemiological Studies Depression Scale (CES-D) is a 20-item self-report scale that measures the severity of depression symptoms over the past week. The scale can be used by individuals between the ages of 6 to 17. Possible range of scores is 0 to 60, with the higher scores indicating the presence of more symptomatology.

SECONDARY OUTCOMES:
Services Assessment for Children and Adolescents - Brief form (SACA) | At enrollment (baseline) and 6 months (study completion)
  The Services Assessment for Children and Adolescents (SACA)-Brief Form gathers data on a child's lifetime and past-year use of 30 service settings, 1 item per setting) that are grouped into four broad areas: inpatient, outpatient, school and other (e.g., mentoring, parent aide, supported work). Response options are Yes, No and Don't Know. Administration time is less than 3 minutes. Higher scores indicate more use of services. Kappa statistics indicated acceptable test-retest reliability.

OTHER OUTCOMES:
Feasibility of Intervention Measure (FIM) | At enrollment (baseline) and 6 months following enrollment
  The The Feasibility of Intervention Measure (FIM) is a 4-item instrument measuring the feasibility on a 5 point scale (Completely Disagree, Disagree, Neither Agree or Disagree, Agree, Completely Agree) of an intervention completed by providers of the intervention. Scores can range from 0-25. A higher mean score indicates higher agreement that intervention is feasible.
Acceptability of Intervention Measure (AIM) | At enrollment (baseline) and 6 months following enrollment
  The Acceptability of Intervention Measure (AIM) is 4-item scale that measures the perception among implementation stakeholders that a given treatment, service, practice, or innovation is agreeable, palatable, and/or satisfactory. Ratings are made on 5-point scale (Completely Disagree, Disagree, Neither Agree or Disagree, Agree, Completely Agree) of an intervention completed by providers of the intervention. Scores can range from 0-25. A higher mean score indicates higher agreement that intervention is feasible.
Intervention Appropriateness Measure (IAM) | At enrollment (baseline) and 6 months following enrollment
  The Intervention Appropriateness Measure (IAM) is 4-item scale that measures the perceived fit, relevance, or compatibility of the innovation or evidence-based practice for a given practice setting, provider, or consumer. Ratings are made on 5-point scale (Completely Disagree, Disagree, Neither Agree or Disagree, Agree, Completely Agree) of an intervention completed by providers of the intervention. Scores can range from 0-25. A higher mean score indicates higher agreement that intervention is appropriate (goodness of fit, suitability, applicability, goodness of match).

CONTACTS AND LOCATIONS:
Overall Officials: Bruno J Anthony, PhD, Principal Investigator — University of Colorado School of Medicine - Anschutz Medical Campus
Locations (1):
- Department of Psychiatry, University of Colorado School of Medicine, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
We will use a dissemination approach to comply with NIH Policy on dissemination of NIH-Funded Clinical Trial Information and to ensure study findings are available to the research and clinical community as well as the general public. Investigators will ensure that clinical trials under the award are registered and results information is submitted to ClinicalTrials.gov as outlined in the NIH Policy on the Dissemination of Clinical Trial Information and according to the specific timelines stated in the Policy. Registration will occur prior to IRB approval but no later than 21 days following enrollment of the first subject. Once a study record is established, required updates will be performed at least once every 12 months,, confirming the completeness and accuracy of the study record. Summary results will be submitted by the standard results submission due date, and any required results updates will be submitted according to ClinicalTrials.gov regulations
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The research resources and data generated from this grant will be freely distributed, as available, to qualified academic investigators for noncommercial research. The data listed above will be uploaded every six months following the onset of data collection (expected date: 3/1/25) to the National Database for Clinical Trials related to Mental Illness after being harmonized to its Data Dictionary. The IDP information (Study Protocol, Statistical Analysis Plan, Informed Consent Form, Clinical Study Report and Analytic Code) will be available 3 months following publication of seminal article of results and ending 5 years following publication.
Access Criteria: Researchers who provide a methodologically sound proposal will have access to the Study Protocol, Statistical Analysis Plan, Informed Consent Form, Clinical Study Report and Analytic Code. Data will be available through the National Database for Clinical Trials. Requests should be sent to Dr. Bruno Anthony (PI) at bruno.anthony@cuanschutz.edu. Data requestors will need to sign a Data Use Agreement.
URL: https://pcmh.org/?x=1xVaO92z

REFERENCES:
- [Background] Pitts BH, Doyle R, Wood L, Dar R, De Jesus Ayala S, Sharma T, St Pierre M, Anthony B. Brief Interventions for Suicidal Youths in Medical Settings: A Meta-Analysis. Pediatrics. 2024 Mar 1;153(3):e2023061881. doi: 10.1542/peds.2023-061881. PMID 38356411
- See also: Site provides access to descriptions of study and relevant background information — https://pcmh.org